CLINICAL TRIAL: NCT07283757
Title: PTSD Treatment for Incarcerated Men and Women: Arnold Ventures (AV)
Brief Title: PTSD Treatment for Incarcerated Men and Women: AV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Arnold Ventures (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-0630: AV; A538900 (Other: UW Madison); Protocol Version 1/23/2026 (Other: UW Madison)
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: PTSD
Keywords: Group therapy; Incarcerated Individuals
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two therapy-intervention groups: CPT or active waitlist control group. Participants will be stratified/randomized based on PTSD severity (PCL-5 total score).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The research members performing the assessments will be blind to the group assignment. One study staff will schedule participants according to the randomization, thus minimizing the possibility of systematically biasing the outcome and mediator assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Processing Therapy (CPT) group (Experimental): Participant groups of 6-10 people to receive CPT to treat PTSD over 6 weeks or 12 weeks, depending on session frequency.
  Interventions: Behavioral: Cognitive Processing Therapy
- Waitlist Control (No Intervention): Participant groups will provide data as a control group first, and will then receive CPT to treat PTSD

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — CPT: a type of cognitive behavioral therapy recommended for the treatment of PTSD. Delivered in 8 - 12, 90-minute sessions with an emphasis on addressing trauma-related cognitions and challenging trauma-related beliefs. Includes homework assignments.
  Arms: Cognitive Processing Therapy (CPT) group

SUMMARY:
This research will help identify if a PTSD treatment group, called Cognitive Processing Therapy (CPT), that is used in community settings is helpful in reducing PTSD symptoms among people who are incarcerated. The goal of CPT is to create a space for people to modify unhelpful beliefs related to trauma. A total of 692 participants will be enrolled from 6 locations and can expects to be on study for up to 24 weeks.

DETAILED DESCRIPTION:
The primary objective of this project is to determine the effectiveness of group CPT in reducing conduct reports (violations of prison rules such assaults and substance use), reducing PTSD symptom severity, and address the long-term outcome of recidivism in male and female incarcerated populations.

Up to 692 incarcerated individuals will participate in group assignment. To account for potential participant attribution between consent, group assignment, and the waitlist group receiving treatment, enrollment could be up to 900 participants. AV branch of the study involves a waitlist control group; this group will receive the CPT treatment after the treatment group completes the treatment. Participation in the waitlist control group will not affect participation in any other treatments that are available at the facilities.

Prior to beginning any study procedures, informed consent will be obtained orally and in writing. During the informed consent process, eligible participants will be provided with detailed information about the study, including their right to refuse or discontinue participation at any time and the fact that their decision to participate or decline will have no bearing on their standing within the criminal justice system.

Potential participants will be contacted by calling them over the phone system within the prison. When they arrive to the private testing room, they are asked if they would like to learn about the study and potentially participate. If so, participants undergo consent.

Eligible participants will complete the PCL-5 to ascertain current PTSD symptomology and probable diagnosis. This assessment will take approximately 90 minutes.

Participants will be randomly assigned to the CPT or the waitlist control group. The CPT group will engage in 8 -12, 90-minute treatment sessions (18 hours total). With the optional opportunity to take 15-20 minutes after each session to de-stress and calm down if necessary. These sessions will take place over 6 to 12 weeks, depending on session frequency. CPT group-members are also asked to complete weekly homework (approximately 12 hours total). A maximum of 10 participants, but no less than 3 will be included in each CPT group. When the waitlist control group reaches the treatment phase, if the participant count fall below 3, additional participants will be enrolled to maintain sufficient numbers. Data collection during treatment will mirror that of the active waitlist control group. Participants will be notified via institutional mail which group they have been enrolled in.

In addition to the treatment groups, CPT and control group members will complete a PCL-5 / PHQ-9 at the beginning of each session. As well as pre-treatment testing session prior to the start of treatment. CPT and control group members will complete post-treatment testing within one week after completing week 6 or 12 of treatment. Facilities will have the option to offer one follow up CPT session 6-12 weeks post-treatment. Final follow-up will occur three months after the end of treatment. Procedures will be the same as other timepoint follow-ups. Participants who receive treatment may be selected for a 1on1 interview to hear about their experiences with the group. CPT and control group members will be asked to complete 15-19 sessions in total (pre-treatment, post- treatment, three-month follow-up treatment, 1on1 interview, 12 group sessions and one optional follow-up CPT session).

ELIGIBILITY:
Participants will be enrolled from the Department of Corrections trauma treatment waitlist who have been screened for:

* No active symptoms of psychosis that would interfere with the individual's ability to participate in the group
* No active suicidal ideation with intent or plan
* Able and willing to participate in group therapy
* 18 years old or older
* meet PCL-5 criteria for current PTSD diagnosis within 2 months of enrollment
* No scheduled release date before the end of the treatment group
* able to understand the consent form as measured by the consent quiz
* have not participated in the previous CPT groups with UW project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Number of Conduct Reports | Up to 26 weeks on study
  Effectiveness of group CPT in reducing conduct reports measured by number of violations of prison rules such assaults and substance use.

SECONDARY OUTCOMES:
Change in PTSD Checklist for DSM-5 (PCL-5) severity score | baseline (pre-intervention), up to 12 weeks (post-intervention), and up to 24 weeks (three months follow up)
  PTSD symptom severity is measured by PCL-5 questionnaire (scores from 0, no symptoms, to 80, high severity). Participants will complete the PCL-5 questionnaire during pre-, post-, and three-month follow up timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Koenigs, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Psychiatric Institute and Clinic, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] James, D.J. and L.E. Glaze, Mental health problems of prison and jail inmates, U.S.D.o. Justice, Editor. 2006: Bureau of Justice Statistics Special Report.
- [Background] Egeressy A, Butler T, Hunter M. 'Traumatisers or traumatised': Trauma experiences and personality characteristics of Australian prisoners. Int J Prison Health. 2009;5(4):212-22. doi: 10.1080/17449200903343209. PMID 25757522
- [Background] Campbell CA, Albert I, Jarrett M, Byrne M, Roberts A, Phillip P, Huddy V, Valmaggia L. Treating Multiple Incident Post-Traumatic Stress Disorder (PTSD) in an Inner City London Prison: The Need for an Evidence Base. Behav Cogn Psychother. 2016 Jan;44(1):112-7. doi: 10.1017/S135246581500003X. Epub 2015 Feb 20. PMID 25697197
- [Background] Resick, P.A., C.M. Monson, and K.M. Chard, Cognitive Processing Therapy for PTSD: A Comprehensive Manual. 2016: Guilford Press.
- [Background] Resick PA, Nishith P, Weaver TL, Astin MC, Feuer CA. A comparison of cognitive-processing therapy with prolonged exposure and a waiting condition for the treatment of chronic posttraumatic stress disorder in female rape victims. J Consult Clin Psychol. 2002 Aug;70(4):867-79. doi: 10.1037//0022-006x.70.4.867. PMID 12182270
- [Background] Morgan RD, Winterowd CL. Interpersonal process-oriented group psychotherapy with offender populations. Int J Offender Ther Comp Criminol. 2002 Aug;46(4):466-82. doi: 10.1177/0306624X02464008. PMID 12150085
- See also: PTSD Treatment for Incarcerated Men and Women: WPP — https://clinicaltrials.gov/study/NCT05432817